CLINICAL TRIAL: NCT06952049
Title: Does Psychoeducation Improve the Pain Relief Derived From a Brief Mindfulness-Based Intervention Delivered in a Clinic Waiting Room
Brief Title: Does Psychoeducation Improve the Pain Relief Derived From a Brief Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004916_PsychoedImpact
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-08

CONDITIONS: Pain; Acute Pain
MeSH Terms: conditions — Pain; Acute Pain | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Pain Psychoeducation (Active Comparator): In the pain psychoeducation intervention, participants will be randomized to listen to a three-minute recording about different pain management strategies (e.g., ice, rest) to promote overall well-being.
  Interventions: Behavioral: Pain Psychoeducation
- Mindfulness without Psychoeducation (Experimental): In the mindfulness without psychoeducation intervention, participants will be randomized to listen to a three-minute mindfulness practice consisting of 1 minute of mindful breathing, 1 minute of mindful mapping, and 1 minute of mindfulness of personal meaning.
  Interventions: Behavioral: Mindfulness without Psychoeducation
- 1 Minute Psychoeducation with 2 Minutes of Mindfulness (Pain Focus) (Experimental): In the 1 Minute Psychoeducation with 2 minutes of Mindfulness (Pain Focus) intervention, participants will be randomized to listen to a 1 minute of psychoeducation about mindfulness, 1 minute of mindful breathing and 1 minute of mindful mapping.
  Interventions: Behavioral: 1 Minute Psychoeducation with 2 Minutes of Mindfulness (Pain Focus)
- 1 Minute Psychoeducation with 2 Minutes of Mindfulness (Meaning Focus) (Experimental): In the 1 Minute Psychoeducation with 2 minutes of Mindfulness (Meaning Focus) intervention, participants will be randomized to listen to a 1 minute of psychoeducation about mindfulness, 1 minute of mindful breathing and 1 minute of mindfulness of personal meaning.
  Interventions: Behavioral: 1 Minute Psychoeducation with 2 Minutes of Mindfulness (Meaning Focus)
- 2 Minutes of Psychoeducation with 1 Minute of Mindfulness (Experimental): In the 2 Minutes of Psychoeducation with 1 Minute of Mindfulness intervention, participants will be randomized to listen to a 2 minute of psychoeducation about mindfulness and 1 minute of mindful breathing.
  Interventions: Behavioral: 2 Minutes of Psychoeducation with 1 Minute of Mindfulness

INTERVENTIONS:
Behavioral: Pain Psychoeducation — In the pain psychoeducation intervention, participants will be randomized to listen to a three-minute recording about different pain management strategies (e.g., ice, rest) to promote overall well-being.
  Arms: Pain Psychoeducation
Behavioral: Mindfulness without Psychoeducation — In the mindfulness without psychoeducation intervention, participants will be randomized to listen to a three-minute mindfulness practice consisting of 1 minute of mindful breathing, 1 minute of mindful mapping, and 1 minute of mindfulness of personal meaning.
  Arms: Mindfulness without Psychoeducation
Behavioral: 1 Minute Psychoeducation with 2 Minutes of Mindfulness (Pain Focus) — In the 1 Minute Psychoeducation with 2 minutes of Mindfulness (Pain Focus) intervention, participants will be randomized to listen to a 1 minute of psychoeducation about mindfulness, 1 minute of mindful breathing and 1 minute of mindful mapping.
  Arms: 1 Minute Psychoeducation with 2 Minutes of Mindfulness (Pain Focus)
Behavioral: 1 Minute Psychoeducation with 2 Minutes of Mindfulness (Meaning Focus) — In the 1 Minute Psychoeducation with 2 minutes of Mindfulness (Meaning Focus) intervention, participants will be randomized to listen to a 1 minute of psychoeducation about mindfulness, 1 minute of mindful breathing and 1 minute of mindfulness of personal meaning.
  Arms: 1 Minute Psychoeducation with 2 Minutes of Mindfulness (Meaning Focus)
Behavioral: 2 Minutes of Psychoeducation with 1 Minute of Mindfulness — In the 2 Minutes of Psychoeducation with 1 Minute of Mindfulness intervention, participants will be randomized to listen to a 2 minute of psychoeducation about mindfulness and 1 minute of mindful breathing.
  Arms: 2 Minutes of Psychoeducation with 1 Minute of Mindfulness

SUMMARY:
This project is a single-site, five-arm, randomized controlled trial investigating whether providing patients in an orthopedic clinic waiting room psychoeducation about mindfulness impacts the degree of pain relief they experience during a mindfulness-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* Receiving pain treatment at Tallahassee Orthopedic Center
* Understanding English instructions fluently
* Being 18 years of age or older

Exclusion Criteria:

* Unable to consent because of physical or mental incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | Immediately before to after 3-minute audio recording
  Change in acute pain unpleasantness will be measured with an individual item ("How unpleasant is your pain, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain unpleasantness.

SECONDARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | Immediately before to after 3-minute audio recording
  Change in acute pain intensity will be measured with an individual item ("How much pain do you have, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain intensity.
Change in Anxiety Numeric Rating Scale | Immediately before to after 3-minute audio recording
  Change in anxiety from baseline will be assessed a single item adapted from the Generalized Anxiety Disorder-2. Scores range from 0 to 10, with higher scores reflecting greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic (TOC), Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No